CLINICAL TRIAL: NCT01988519
Title: Does the Type of Drain Influence the Postoperative Pancreatic Fistula Rate After Pancreatic Resection?
Brief Title: Randomized Controlled Trial Comparing Closed-suction Drain Versus Passive Gravity Drain Following Pancreatic Resection
Acronym: DRAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Filip Cecka, MUDr. Filip Čečka, Ph.D., University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNHK 13
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Pancreaticoduodenectomy; Distal Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed suction drain (Active Comparator): Two closed suctions drains will be placed near the pancreatic anastomosis or suture line. The drains will be removed on the 4th or 5th day if the amylase activity is not increased.
  Interventions: Procedure: closed suction drain
- Closed gravity drain (Active Comparator): Two closed gravity drains will be placed near the pancreatic anastomosis or suture line. The drains will be removed on the 4th or 5th day if the amylase activity is not increased.
  Interventions: Procedure: Closed gravity drain

INTERVENTIONS:
Procedure: Closed gravity drain — passive tube drains (PFM Medical, Köln, Germany)
  Arms: Closed gravity drain
Procedure: closed suction drain — BLAKE Silicon drains (Ethicon, USA)
  Arms: Closed suction drain

SUMMARY:
Pancreatic resection is the only potentially curative modality of treatment for pancreatic neoplasm. The mortality associated with this procedure decreased rapidly in the past decades. However, the morbidity associated with pancreatic resection remains high. The main reason for postoperative morbidity is postoperative pancreatic fistula (POPF), which is regarded as the most ominous complication following pancreatic resection. Its reported incidence varies in the surgical literature from 10% to >30%.

Recently published studies showed that the placement of intraoperative drains, manipulation with the drains, timing of removal of the drain, and especially the type of drain, have significant effect on the postoperative complications, and especially POPF.

Controversy exists regarding the type of intraoperatively placed drain. Nowadays, the two most commonly used systems are closed suction drainage and closed gravity drainage. Open systems have been abandoned in most centers as they are obsolete.

Our hypothesis is that the closed suction drain will have better results as it is more effective than the gravity drainage. However, some surgeons claim that the suction system can actively suck the pancreatic juice through the anastomosis or suture and thus promote the development of POPF.

The aim of this study is to compare closed suction drains and closed gravity drains after pancreatic resection in a randomized controlled study.

The primary end-point is the postoperative pancreatic fistula rate. The secondary end-point is the postoperative morbidity.

DETAILED DESCRIPTION:
Pancreatic resection is the only potentially curative modality of treatment for pancreatic neoplasm. The mortality associated with this procedure decreased rapidly in the past decades. However, the morbidity associated with pancreatic resection remains high. The main reason for postoperative morbidity is postoperative pancreatic fistula, which is regarded as the most ominous complication following pancreatic resection. Its reported incidence varies in the surgical literature from 10% to >30%.

Recently published studies showed that the placement of intraoperative drains, manipulation with the drains, timing of removal of the drain, and especially the type of drain, have significant effect on the postoperative complications, and especially POPF.

Even though several trials showed that the routine use of intraoperatively placed drains in elective pancreatectomy does not reduce postoperative morbidity, most of the high-volume pancreatic surgery centers still place the drains routinely. The theoretical advantage of drainage is to identify an early bile or pancreatic leak, or postoperative hemorrhage; and therefore allow for early treatment of the complication; or in some cases, the drain would control the leak without necessity of reintervention.

Two large studies compared early versus late removal of the intraoperatively placed drains. The first published by Kawai et al. was a cohort study, including 104 patients. The second one published by Bassi et al. was prospective randomized trial including 114 patients. Both studies clearly showed that the group of patients with early drain removal has superior results, lower rate of POPF and lower morbidity.

Controversy exists regarding the type of intraoperatively placed drain. The surgeons in the USA usually use the closed suction drainage system. On the other hand, European and Asian surgeons usually prefer open Penrose system, closed gravity drainage, or a combination of both. The closed suction drainage system uses slight under pressure to drain the fluid from the abdominal cavity. It is more effective than other systems, and thus advantageous. However, some surgeons claim that the suction system can actively suck the pancreatic juice through the anastomosis or suture and thus promote the development of POPF.

Only one study published by Schmidt et al. compared closed suction drainage system with gravity drainage. However, this study collected results over a very long period, and the comparison of the drains was not primary end-point of the study. Randomized controlled trials comparing various drains were published in cardiac surgery.

The situation in pancreatic surgery is specific. The pancreatic anastomosis or suture line is not water-tight in large proportion of cases. It is due to the character of pancreatic parenchyma. Especially in soft pancreas, the stitches can cut through and cause leak of the suture line or anastomosis. Therefore, pancreatic leak is not rare after pancreatic resections. Most of the POPF are grade A according to the ISGPF classification; with no clinical consequences. The aim of the postoperative management should prevent the POPF become clinically more severe (grade B and C). And the manipulation with the drains, and especially the type of drain, seem to play a major role.

ELIGIBILITY:
Inclusion Criteria:

* pancreaticoduodenectomy
* distal pancreatectomy

Exclusion Criteria:

* central pancreatectomy
* total pancreatectomy
* enucleation
* laparoscopic procedure
* resection and reconstruction of portal vein

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula | 30 days postoperatively
  Postoperative pancreatic fistula defined according to the ISGPF (International Study Group for Pancreatic Fistula)

SECONDARY OUTCOMES:
Postoperative morbidity | 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Filip Cecka, MD, PhD, Principal Investigator — Department of Surgery, University Hospital Hradec Kralove
Locations (2):
- Czechia (2):
  - Department of Surgery, Hradec Králové
  - Department of Surgery, Olomouc

REFERENCES:
- [Background] Cecka F, Lovecek M, Jon B, Skalicky P, Subrt Z, Ferko A. DRAPA trial--closed-suction drains versus closed gravity drains in pancreatic surgery: study protocol for a randomized controlled trial. Trials. 2015 May 7;16:207. doi: 10.1186/s13063-015-0706-1. PMID 25947117